CLINICAL TRIAL: NCT04618718
Title: Cerebral Protection in Transcatheter Aortic Valve Replacement - The PROTEMBO C Trial
Brief Title: The PROTEMBO C Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protembis GmbH (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP_00105
Record Dates: First submitted 2020-10-20; First posted 2020-11-06 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Valvular Heart Disease
Keywords: TAVR; cerebral embolic protection
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): ProtEmbo device will be used as distal protection device in subjects undergoing TAVR
  Interventions: Device: cerebral embolic protection during TAVR

INTERVENTIONS:
Device: cerebral embolic protection during TAVR — The ProtEmbo system is an adjunctive device placed in the central arterial system at the beginning of a TAVR procedure to deflect embolic particles during the procedure and removed following the completion of the procedure.

SUMMARY:
The PROTEMBO C Trial is an international, multi-center, single arm, non-inferiority study of the safety and performance of using the ProtEmbo System for cerebral embolic protection in subjects with severe native aortic valve stenosis indicated for TAVR.

ELIGIBILITY:
Inclusion Criteria:

1. The heart team recommends transcatheter valve aortic valve replace consistent with the 2017 ESC/EACTS Guidelines for the management of valvular heart disease.
2. Compatible left subclavian artery (≥ 4 mm diameter) without significant stenosis (> 70%) and distance between the origin of left subclavian artery and valve plain of ≥ 90mm as determined by Multi-Slice Computed Tomography (MSCT) scan or equivalent imaging modality.
3. The subject and the treating physician agree that the subject will undergo the scheduled pre-procedural testing and return for all required post-procedure follow-up visits.
4. The subject is able to provide informed consent, has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the relevant regulatory authority of the respective clinical site.
5. Subject is a minimum of 18 years of age.

Exclusion Criteria:

General:

1. Left upper limb vasculature in the left extremity precluding 6Fr sheath radial / brachial / subclavian access.
2. Inadequate circulation to the left extremity as evidenced by signs of artery occlusion (modified Allen's test) or absence of radial/brachial pulse.
3. Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature.
4. TAVR conducted via other than transfemoral access (subclavian, axillar, transapical, transaortic, carotid or transcaval).
5. Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment.
6. Aortic valve is a congenital unicuspid or bicuspid valve.
7. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
8. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease).
9. Blood dyscrasias as defined: Leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy.
10. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
11. Need for emergency surgery for any reason.
12. Severe hypertrophic cardiomyopathy with or without obstruction.
13. Severe ventricular dysfunction with LVEF ≤30%.
14. Echocardiographic evidence of intracardiac or aortic mass, thrombus, or vegetation.
15. Symptomatic or asymptomatic severe (≥ 70%) occlusive carotid disease requiring concomitant CEA / stenting.
16. Subject has undergone carotid stenting or carotid endarterectomy within the previous 6 weeks.
17. Active peptic ulcer or upper GI bleeding within the prior 6 months.
18. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, or clopidogrel, device component material, or sensitivity to contrast media, which cannot be adequately premedicated.
19. Recent (within 6 months) CVA or a TIA.
20. Renal insufficiency (creatinine > 3.0 mg / dL or GFR < 30) and / or renal replacement therapy at the time of screening.
21. Life expectancy < 12 months due to non-cardiac co-morbid conditions.
22. Subjects in whom anti-platelet and / or anticoagulant therapy is contraindicated, or who will refuse transfusion.
23. Subjects who have active bacterial endocarditis or other active infections.
24. Currently participating in an investigational drug or another device study.
25. Subjects who have a planned treatment with any other investigational device or procedure during the study follow-up period (30 days).
26. Subjects with planned concomitant surgical or transcatheter ablation for Atrial Fibrillation during the study follow-up period (30 days).
27. Any subject with a balloon valvuloplasty (BAV) within 30 days of the procedure.
28. Subject is a woman of child-bearing potential.
29. Patient with Heparin-Induced Thrombocytopenia Syndrome.
30. Inner diameter of aortic arch is less than 25mm.
31. Brachiocephalic trunk originating from the aortic arch that splits into the bilateral subclavian arteries and a bicarotid trunk (Origin D).
32. Hepatic failure (defined as liver enzyme elevations two times the upper limit of normal) or active infectious hepatitis
33. Cardiogenic shock or severe hypotension (systolic blood pressure < 90 mm Hg) at the time of the index procedure
34. Subjects who have a planned concomitant cardiac surgical or interventional procedure (e.g., coronary revascularization) during the TAVI procedure
35. Subjects who have a pre-existing prosthetic heart valve in any position

Neurological:

1. Subject had active major psychiatric disease.
2. Subject has severe visual, auditory, or learning impairment and is unable to comprehend English or local language and therefore unable to be consented for the study.
3. Subjects with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Angiographic:

1. Excessive tortuosity or severe peripheral arterial disease in the left radial / brachial / subclavian artery preventing ProtEmbo System access and insertion.
2. Subject whose left radial / brachial / subclavian artery reveals significant stenosis, calcification, ectasia, dissection, occlusion or aneurysm, in particular at or within 3 cm of the aortic ostium.
3. Subject with significant stenosis, ectasia, dissection, or aneurysm in the ascending aorta or in the aortic arch, or with abnormal aortic arch angulation or abnormal anatomical conditions of the aorta.

Magnetic Resonance Imaging:

1. Subject Body Mass Index (BMI) precluding imaging in scanner.
2. Contraindications to MRI (subjects with any implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure).
3. Subjects who have a high risk of complete AV block after TAVR, with the need of permanent pacemaker (e.g. subjects with preexisting bifascicular block or complete right bundle branch block plus any degree of AV block).
4. Planned implantation of a pacemaker or defibrillator implantation within the first 4 days after TAVR.
5. Claustrophobia precluding MRI scanning.
6. No scanner hardware, software, coil or protocol changes during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (4):
  - Krankenhaus der Barmherzigen Brüder Trier, Trier, Rhineland-Palatinate
  - Herzzentrum Leipzig-Universitätsklinik für Kardiologie-Helios, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein (UKSH), Lübeck, Schleswig-Holstein
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny Przemienienia Panskiego Poznan University of Medical Sciences, Poznan
  - Department of Interventional Cardiology Warsaw Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fezzi S, Jagielak D, Targonski R, Schmidt T, Frerker C, Witkowski AR, Lauterbach M, Leick J, Erglis A, Narbute I, Grygier M, Misterski M, Frank D, Abdel-Wahab M, Wilde J, Adam M, Gatto F, Zivadinov R, Dwyer M, Werner N, Mylotte D. Final report of the PROTEMBO C Trial: a prospective evaluation of a novel cerebral protection device during TAVI. EuroIntervention. 2024 Feb 19;20(4):e264-e267. doi: 10.4244/EIJ-D-23-00743. No abstract available. PMID 38389472
- [Result] Jagielak D, Targonski R, Frerker C, Abdel-Wahab M, Wilde J, Werner N, Lauterbach M, Leick J, Grygier M, Misterski M, Erglis A, Narbute I, Witkowski AR, Adam M, Frank D, Gatto F, Schmidt T, Lansky AJ. Safety and performance of a novel cerebral embolic protection device for transcatheter aortic valve implantation: the PROTEMBO C Trial. EuroIntervention. 2022 Sep 20;18(7):590-597. doi: 10.4244/EIJ-D-22-00238. PMID 35608032

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: ProtEmbo device will be used as distal protection device in subjects undergoing TAVR cerebral embolic protection during TAVR: The ProtEmbo system is an adjunctive device placed in the central arterial system at the beginning of a TAVR procedure to deflect embolic particles during the procedure and removed following the completion of the procedure.
Period: Overall Study
Arm/Group | Intervention
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 5
  Poland | 39
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participants With MACCE Events
Description: Number of participants experiencing a Major Adverse Cardiac and Cerebrovascular Event (MACCE) defined by VARC-2 including all-cause mortality, all stroke, life-threatening or disabling bleeding, vascular injury and acute kidney injury (stage 2 or 3) within 30 days of the procedure
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 64
Participants | 3

2. Primary Outcome: Rate of Participants in Whom Technical Success Was Achieved
Description: Number of participants in whom technical success was achieved during the procedure. Technical success is defined as the ability to safely deliver, deploy, and remove the device, ability to secure positioning and stability of the position throughout the transcatheter intracardiac procedure and ability to deflect embolic material as assessed by adequate coverage while not impeding blood flow, deployed and removed and positioning and stability of the device
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
Participants | 57

3. Secondary Outcome: Efficacy-MR Imaging: Comparison Between the Median New Lesion Volume in the Brain
Description: Comparison between the median new lesion volume in the brain assessed by diffusion weighted magnetic resonance images (DW-MRI) at 2-7 days and historical data; the total new lesion volume is defined as the sum of all diffusion-positive new cerebral lesions in post-procedural DW-MRI relative to the pre-TAVR DW-MRI
Time Frame: 2-7 days post-procedure
Measure: Median (Inter-Quartile Range); unit: mm3
Arm/Group | Intervention
Number analyzed (Participants) | 51
mm3 | 210 [108 to 566]

4. Secondary Outcome: Composite Rate of Death or All Strokes
Description: Death or all stroke according to VARC-2 criteria (to define occurrence and type stroke) within 3 days (72 hours) of the TAVR procedure compared to historical data
Time Frame: 3 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 64
Participants | 1

ADVERSE EVENTS:
Time Frame: 30 days (+/- 7 days)
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 20/64
Other Adverse Events (participants affected / at risk) | 21/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=64)
Drop in Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
1st degree AV Block (Cardiac disorders) | 1 (1)
3rd degree AV block (Cardiac disorders) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1)
Left Bundle Branch Block (Cardiac disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Tamponade/Sternotomy (Surgical and medical procedures) | 1 (1)
Radial artery dissection (Surgical and medical procedures) | 1 (1)
Sedative Circulatory Complication (Surgical and medical procedures) | 1 (1)
TAVR access site complication (Surgical and medical procedures) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=64)
Abnormal Alkaline Phosphatase and Gamma GT (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Left Anterior Fascicular Block (Cardiac disorders) | 1 (1)
Left Bundle Branch Block (Cardiac disorders) | 2 (2)
Diarrhea (Infections and infestations) | 1 (1)
Loss of Sphincter Tone (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Radial Artery Occlusion (Surgical and medical procedures) | 2 (2)
Postoperative nausea and vomitting/ vertigo (Surgical and medical procedures) | 1 (1)
Short period of delirium post TAVR (Nervous system disorders) | 1 (1)
TAVR access site hematoma (Vascular disorders) | 2 (2)
Vascular access site hematoma (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT04618718/Prot_SAP_000.pdf